CLINICAL TRIAL: NCT06936059
Title: A Prospective, Randomized, Parallel-controlled Clinical Trial to Evaluate the Effectiveness and Safety of Chronic Pain Rehabilitation Training Software in Assisting in the Relief of Chronic Secondary Musculoskeletal Pain
Brief Title: A PRPCT to Assess the Efficacy & Safety of Chronic Pain Rehab Training Software for Alleviating Chronic Secondary Musculoskeletal Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: XH-24-010
Record Dates: First submitted 2025-01-23; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain
Keywords: pain; Visual Pain Score; rehab training software; anxious; depressed
MeSH Terms: conditions — Chronic Pain; Pain; Anxiety Disorders; Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Change in pain intensity before and after MR therapy (Experimental): A 30% decrease in VAS score compared to the screening period is valid
  Interventions: Device: Mixed Reality based analgesic therapy
- Placebo version of chronic pain rehabilitation training software (Placebo Comparator): We use the same non-mixed reality（Non-MR） scenario to treat patients, although the scenario is completely identical, it is not presented in a mixed reality scenario.
  Interventions: Device: Mixed Reality based analgesic therapy

INTERVENTIONS:
Device: Mixed Reality based analgesic therapy — The intervention is a single 15 min MR therapy. The MR therapy is consisted of MR device and software. The model of MR device used is Pico Neo 3 Pro. The software run on the MR device delivers two types of contents: 1) A 7min of computer-generated 360 video of underwater scene with therapeutic music to distract patients' attention on pain and make patients passively relax. 2) An 8min guided relaxation in which patients are transported to seaside with narrative to achieve image and breathing relaxation.
  And the placebo-group used the same non-mixed reality(Non-MR) scenario to treat patients, although the scenario is completely identical, it is not presented in a mixed reality scenario. It only presents the scene in normal display mode.

SUMMARY:
A prospective, randomized, parallel-controlled clinical trial to evaluate the effectiveness and safety of chronic pain rehabilitation training software in assisting in the relief of chronic secondary musculoskeletal pain

DETAILED DESCRIPTION:
A PRPCT to assess the efficacy & safety of chronic pain rehab training software for alleviating chronic secondary musculoskeletal pain

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥18 years old.
* Average pain intensity≥4 on a 0-10 numerical rating scale (NRS) in the past 24 hours.
* Be able to communicate in Chinese.
* Be able to read and write Chinese.
* Willing to comply with study procedures and restrictions.
* Willing and able to sign informed consent.

Exclusion Criteria:

* Shingles on the eyes, ears, head, face, or hands.
* Trigeminal neuralgia.
* Severe vision impairment. (Patients with clear vision wearing glasses or contact lenses are allowed)
* Severe hearing impairment.
* Disease or medical condition predisposing to nausea or dizziness, such as insufficient blood supply to the brain, vestibular dysfunction,cholecystitis, etc.
* History of severe motion sickness.
* Injury to eyes, ears, face, or neck that impedes comfortable use of mixed reality.
* Injury or dysfunction of hands or upper limbs that impedes comfortable use of mixed reality.
* Diagnosis of cognitive impairment, epilepsy, dementia, migraines or other neurological diseases that may prevent the use of mixed reality.
* History of mental illness, including depression, generalized anxiety disorder, schizophrenia, etc.
* Females currently pregnant.
* Current or completion of participation within 4 weeks before screening in any interventional clinical study
* Patients whom the investigator considers not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-12 (Estimated); Primary Completion 2026-11-12 (Estimated); Study Completion 2026-11-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity before and after MR therapy | 20min
  The pain intensity is measured using a 0-10 numerical rating scale (NRS) of pain. The anchors for the numerical rating scale were "Ten is the worst pain anyone could ever have and zero is no pain at all." Before the MR therapy started, the participant would be asked what his or her pain level is on the 0-10 numerical rating scale. After the 15 minute MR therapy, the participant would be asked what his or her pain level at that moment, again using the 0-10 numerical rating scale. The change in pain intensity before and after MR therapy is then obtained with the two pain level numbers subtracted.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua hospital ,Shanghai Jiaotong University, School of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
To protect the personal information privacy of participants